CLINICAL TRIAL: NCT04100460
Title: A Randomized, Placebo-controlled, Crossover Study to Investigate the Effect of Arabinoxylan on Gastrointestinal Tolerance and Microbial Changes in Generally Healthy Adults.
Brief Title: A Double Blind Study on the Gastrointestinal Effects of Arabinoxylan (Leaf Fiber Extract).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Comet Bio Inc. (Industry)
Collaborators: Biofortis, Merieux NutriSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BIO-1907
Record Dates: First submitted 2019-09-12; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Tolerance
Keywords: Fecal Microbiota; Gastrointestinal tolerance; Bowel habits

STUDY DESIGN:
Intervention Model Description: The study is a randomized, placebo-controlled, crossover, singe-center trial with one screening visit and 3 test periods separated by minimum 2 - week washout periods.
Who Masked: Participant, Investigator
Masking Description: Study personnel will remain blinded to the sequence assigned to subjects throughout the study. A set of sealed unblinding envelopes will be provided to the Clinical Investigator for use in an emergency situation where a subject's health is at risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 7.25 grams of Arabinoxylan leaf fiber extract (Experimental): Participants are given 7.25 grams of Arabinoxylan daily
  Interventions: Dietary Supplement: 7.25 grams of Arabinoxylan leaf fiber extract
- 14.5 grams of Arabinoxylan leaf fiber extract (Experimental): Participants are given 14.5 grams of Arabinoxylan daily
  Interventions: Dietary Supplement: 14.5 grams of Arabinoxylan leaf fiber extract
- Control - No Arabinoxylan (Maltodextrin) (Placebo Comparator): Participants are given no Arabinoxylan
  Interventions: Dietary Supplement: Control - No Arabinoxylan

INTERVENTIONS:
Dietary Supplement: 7.25 grams of Arabinoxylan leaf fiber extract — Participants are given 7.25 grams of Arabinoxylan daily
  Arms: 7.25 grams of Arabinoxylan leaf fiber extract
Dietary Supplement: 14.5 grams of Arabinoxylan leaf fiber extract — Participants are given 14.5 grams of Arabinoxylan daily
  Arms: 14.5 grams of Arabinoxylan leaf fiber extract
Dietary Supplement: Control - No Arabinoxylan — Participants are given no Arabinoxylan
  Arms: Control - No Arabinoxylan (Maltodextrin)

SUMMARY:
The objective of this study is to investigate the effect on Arabinoxylan on gastrointestinal (GI) tolerance, bowel habits, and microbiota in adults. The study is a randomized, placebo-controlled, crossover, single-center trial with 3 study periods separated by minimum 2-week washout periods. 45 healthy adults will be recruited for the trial. Participants will be required to drink a beverage twice a day for 3 weeks during each study period. The beverage will contain either approximately 7.25 grams of Arabinoxylan leaf fiber extract per day, or approximately 14.5 grams of Arabinoxylan leaf fiber extract per day, or will not contain any Arabinoxylan (control). Subjects will record their bowel movements daily, fill out daily questionnaires about their gastrointestinal systems, and record their food intake at specified times during the study. Stool samples will also be collected prior to and at the end of each study period for analysis of bacteria composition.

DETAILED DESCRIPTION:
The study is a randomized, placebo-controlled, crossover, single-center trial with one screening visit (Visit 1; Week -1) and 3 test periods [Test Period 1 (Visits 2 and 3; Weeks 0 to 3), Test Period 2 (Visits 4 and 5; Weeks 5 to 8), and Test Period 3 (Visits 6 and 7; Weeks 10 to 13)] separated by minimum 2-week washout periods.

At Visit 1 (Week -1), subjects will provide informed consent and undergo assessments of medical history and prior, current medication/supplement use, and inclusion and exclusion criteria and a last menses query, where applicable. Additionally, height, body weight, and vital signs will be measured and BMI will be calculated. Fasting (12 ± 2 h) blood samples will be collected for chemistry and hematology, and female subjects will undergo an in-clinic urine pregnancy test. Subjects will be instructed to maintain physical activity and habitual diet as much as possible with the exception of excluding fermented foods or beverages that do or might contain live probiotics (e.g., yogurt, kombucha). Subjects will be dispensed a Baseline Diet Diary with instructions to record intake 7 days prior to Visit 2 (Week 0). Subjects will also be dispensed a Bowel Habits Diary and Daily GI Tolerance Questionnaire with instructions to complete these during the 7 days prior to Visit 2 (Week 0). Finally, subjects will be dispensed a stool collection kit and will be instructed to collect one fecal sample from one bowel movement during the 3 days prior to Visit 2 (Week 0). Subjects will be reminded that they are not required to fast prior to Visit 2 (Week 0) and will be encouraged to eat breakfast prior to their visit.

At Visit 2 (Week 0), subjects will arrive at the clinic to undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight and vital signs measurements, last menses query, where applicable). Subjects will be queried about compliance with study instructions. The fecal sample will be collected and the Bowel Habits Diary, Baseline Diet Diary, and Daily GI Tolerance Questionnaire will be collected and reviewed. Subjects will be assigned to a randomization sequence. The first study product consumption will occur in the clinic and subject will be dispensed the remaining study products according to their assigned randomization sequence for home consumption (twice a day, once in the morning and once in the evening, with or without food). Subjects who consumed breakfast at home prior to arriving at the clinic will be administered the study product alone while those who did not consume breakfast prior to arriving at the clinic will be administered the study product with a snack. Subjects will also be dispensed a Study Product Diary to record study product intake. Subjects will be dispensed a copy of the last 5 days of their completed Baseline Diet Diary (reviewed at Visit 2, Week 0) and will be instructed to replicate the same food and beverage intake as closely as possible during the days prior to the collection of their fecal sample, which will occur during the 3 days immediately prior to Visit 3 (Week 3). Additionally, subjects will be dispensed 3-day Analysis Diet Records with instructions to record all food and beverages consumed during 3 days (2 weekdays and one weekend) following Visit 2 (Week 0) and before Visit 3 (Week 3) that do not coincide with the 5 replication days immediately prior to Visit 3 (Week 3). Subjects will be dispensed a Bowel Habits Diary and stool collection kit, and will be instructed to complete the Bowel Habits Diary during the 7 days immediately prior to Visit 3 (Week 3) and to collect a fecal sample from one bowel movement during the 3 days immediately prior to Visit 3 (Week 3). Subjects will also be dispensed a Daily GI Tolerance Questionnaire with instructions to complete the questionnaire daily starting from Visit 2 (Week 0) up to Visit 3 (Week 3). Finally, study instructions will also be provided [(i.e., overnight fasting (12 ± 2 h, water only), maintenance of physical activity with the exception of avoiding vigorous physical activity for 24 h prior; maintenance of habitual diet as much as possible with the exception of avoiding alcohol for 24 h prior and excluding fermented foods or beverages that do or might contain live probiotics (e.g., yogurt, kombucha) and consumption of study products].

At Visit 3 (Week 3), subjects will arrive at the clinic to undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight, and vital signs measurements, last menses query, where applicable) and adverse event (AE) assessments. Subjects will be queried about compliance with study instructions and diet replication. Fasting (12 ± 2 h) blood samples will be collected for chemistry and hematology. Fecal samples will be collected and the Bowel Habits Diary, Daily GI Tolerance Questionnaire, and the 3-day Analysis Diet Record will be collected and reviewed. The Study Product Diary will be collected/reviewed, any unused study products will be collected, and compliance with study product consumption will be assessed. The Product Likeability Questionnaire will be administered in clinic. Subjects will be dispensed a stool collection kit and will be instructed to collect a fecal sample from one bowel movement during the 3 days immediately prior to Visit 4 (Week 5). Subjects will also be dispensed a copy of the last 5 days of their completed Baseline Diet Diary (reviewed at Visit 2, Week 0) and will be instructed to replicate the same food and beverage intake as closely as possible during the days prior to the collection of their fecal sample, which will occur during the 3 days immediately prior to Visit 4 (Week 5). Subjects will also be instructed to begin the 2-week washout period and return to the clinic to begin Test Period 2 at Visit 4 (Week 5). Finally, study instructions will also be provided [(i.e., maintenance of physical activity; maintenance of habitual diet as much as possible with the exception of excluding fermented foods or beverages that do or might contain live probiotics (e.g., yogurt, kombucha)]. Subjects will also be reminded that they are not required to fast prior to Visit 4 (Week 5) and will be encouraged to eat breakfast prior to their visit.

At Visit 4 (Week 5), subjects will return to the clinic, crossover to the other study product in their test sequence, and repeat the procedures from Visits 2 (Week 0) with the exception of the randomization procedure. At Visit 5 (Week 8), subjects will repeat the procedures from Visit 3 (Week 3), followed by a 2-week washout period before starting Test Period 3 at Visit 6 (Week 10). At Visit 6 (Week 10), subjects will return to the clinic, crossover to the other study product in their test sequence, and repeat the procedures from Visits 2 (Week 0) with the exception of the randomization procedure. Finally, at Visit 7 (Week 13), subjects will repeat the procedures from Visit 3 (Week 3).

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18.5 to 35.0 kg/m2 at Visit 1
* Non- smokers/former users (cessation less than or equal to 12 months)
* Regular bowel movements; not constipated
* Willing to maintain physical activity patterns, body weight, and habitual diet throughout the trial
* Willing to limit alcohol consumption to less than or equal to 2 drinks per day
* Willing to avoid vigorous physical activity for 24 hrs prior to and during visits
* Willing to refrain for exclusionary medications, supplements, and products throughout study.
* Willing to comply with the visit schedule and fecal sample collection/processing/storage requirements
* No health conditions that would prevent him/her from fulfilling the study requirements based on medical history and routine laboratory test results.
* Understands the study procedures and signs forms providing consent and authorization of release of relevant protected health information to investigator

Exclusion Criteria:

* Abnormal laboratory test results of clinical significance at Visit 1
* Clinically important GI condition that would potentially interfere with the evaluation of the study product
* Recent (within 2 weeks of Visit 1) history of an episode of acute GI illness
* Self reported history (within 6 weeks of visit 1) of constipation
* Uncontrolled and/or clinically important pulmonary, cardiac, hepatic, renal, endocrine, hematologic, immunologic, neurologic, psychiatric or biliary disorders
* Uncontrolled hypertension
* Known allergy, intolerances or sensitivity to any of the ingredients in the study product
* Extreme dietary habits
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer
* Major trauma or any other surgical event within 3 months of Visit 1
* Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1
* Weight loss or gain of greater than 4.5 kg in the 3 months prior to Visit 1
* Currently or planning to be on a weight loss regimen during the duration of the study
* Antibiotic use within 3 months of Visit 1
* Use of steroids within 1 month of Visit 1
* Chronic use of anti-inflammatory medications within 1 month of Visit 1
* Use of medications and or dietary supplements known to influence GI function
* Consumption of fermented foods or beverages that do or might contain live probiotics within 2 weeks of Visit 1
* Participated in endoscopy or endoscopy prep within 3 months of Visit 1
* Female that is pregnant, planning to be pregnant during the study period, lactating, or is unwilling to use a medically approved form of birth control during the study period
* Recent history (within 12 months of screening) of substance abuse
* Has a condition the Investigator believes will interfere with the subjects inability to provide informed consent, confound the interpretation of the results, or put the subject at risk

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
GI Symptoms Score | 3 weeks +/- 3 days
  Composite GI symptoms Scores obtained from the Daily GI Tolerance Questionnaire will be obtained by summing the ratings to the 8 individual scores (see below in Outcome 2).
Individual GI symptoms ratings | 3 weeks +/- 3 days
  Ratings for each of the 8 individual GI symptoms Scores [gas/flatulence, nausea, vomiting, abdominal cramping, abdominal distention/bloating, borborygmus/stomach rumbling, burping, and/or reflux (heartburn)] will be ranked on a 4-point scale (none, mild, moderate, severe) for symptoms experienced over the previous 24 hours.

SECONDARY OUTCOMES:
Bowel Habits Dairy | 3 weeks +/- 3 days
  Compilation of bowel habits obtained by each subject's Bowel Habits Diary
Fecal Microbiome | 3 weeks +/- 3 days
  Results of the stool samples that will examine diversity, composition, and changes in bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — Biofortis, Merieux NutriSciences; Rich Troyer, Study Director — Comet Bio Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- See also: What we eat in America, NHanes 2015-2016 — http://www.ars.usda.gov/ARSUserFiles/80400530/pdf/1516/Table_1_NIN_GEN_15.pdf